CLINICAL TRIAL: NCT07310966
Title: Comparison of Lithotomy Versus Lateral Position in Retrograde Intrarenal Surgery for Lower Calyceal Stones Less Than 2 cm: A Randomized Controlled Trial
Brief Title: Comparison of Lithotomy Versus Lateral Position in Retrograde Intrarenal Surgery for Lower Calyceal Stones Less Than 2 cm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ammar Fathi Mohamed AlOrabi, Dr, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Patient position in RIRS
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Renal Calculi
Keywords: lithotomy position; lateral position; lower calyx; FURS; RIRS
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithotomy position group (Active Comparator): patients of this group undergo RIRS in Lithotomy position
  Interventions: Procedure: Lithotomy Position
- Lateral position group (Active Comparator): patients of this group undergo RIRS in lateral position
  Interventions: Procedure: Lateral position

INTERVENTIONS:
Procedure: Lithotomy Position — Patients undergo RIRS in lithotomy position
  Arms: Lithotomy position group
Procedure: Lateral position — Patients undergo RIRS in lateral position
  Arms: Lateral position group

SUMMARY:
Retrograde intrarenal surgery (RIRS) is an established minimally invasive treatment for renal stones, particularly for lower calyceal stones less than 2 cm, offering acceptable stone-free rates with low morbidity.

However, stone clearance in the lower calyx remains technically challenging due to unfavorable anatomy, limited scope deflection, and gravity-dependent fragment retention. Patient positioning during RIRS has been suggested as a modifiable factor that may influence endoscopic access, stone relocation, and surgical ergonomics.

The lithotomy position is conventionally used during RIRS, while the lateral position has been proposed to facilitate stone migration and improve lower calyceal access through gravitational assistance. Existing studies comparing patient positioning during RIRS are limited, with most evidence derived from retrospective analyses or non-randomized designs.

Therefore, this randomized controlled trial aims to compare lithotomy versus lateral positioning during RIRS for lower calyceal stones less than 2 cm in terms of operative and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Single or multiple lower calyceal renal stones with stone size <2 cm confirmed by NCCT.
* Negative urine culture.
* Presented cases.

Exclusion Criteria:

* Multiple stones involving renal pelvis or other calyces.
* Anatomical anomalies affecting ureteroscope access (horseshoe kidney, malrotation, ureteral strictures).
* Pregnancy.
* Prior ipsilateral renal surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Stone Free Rate | 1 month
  Stone-free rate (SFR), defined as no clinically significant residual stones on non-contrast 3-mm-cuts CT, measured as yes or no

SECONDARY OUTCOMES:
Operative time | The operative time
  operative time is defined as time between starting the procedure and termination of it measured in minutes
Complications | 1 month
  Intra and postoperative complications, defined as complications happens intraoperative and postoperatively, graded by modified clavien-dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shebin El-Kom, Menoufia, Egypt